CLINICAL TRIAL: NCT02078479
Title: Repetitive Transcranial Magnetic Stimulation in Neuropathic Pain Secondary to Malignancy.
Brief Title: rTMS as a Treatment of Neuropathic Pain Secondary to Malignancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman M. Khedr, Clinical Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rTMS with malignancy pain
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-02

CONDITIONS: Malignancy
Keywords: Malignancy; VAS; LANSS; VDS; Neuropathic pain; rTMS; motor cortex; analgesia
MeSH Terms: conditions — Neoplasms; Neuralgia; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real rTMS (Active Comparator): The active group received Real rTMS over the hand area of motor cortex (20 Hz, 10 second, 10 trains with inter-train interval 30 second with total pulses 2000, intensity 80% of motor threshold) every day for ten consecutive days (5 days/week).
  Interventions: Procedure: 20 Hz, 10 s, 10 trains with inter-train interval 30 s 2000 pulses , intensity 80% over hand area daily for 10 consecutive days (5 days/week).
- Sham rTMS (Sham Comparator): Sham-rTMS was applied using the same parameters but with the coil elevated and angled away from the head to reproduce the same of subjective sensation of rTMS
  Interventions: Procedure: sham rTMS (same parameters but with coil elevated and angled away from the head)every day for ten consecutive days (5 days/week).

INTERVENTIONS:
Procedure: 20 Hz, 10 s, 10 trains with inter-train interval 30 s 2000 pulses , intensity 80% over hand area daily for 10 consecutive days (5 days/week).
  Arms: Real rTMS
Procedure: sham rTMS (same parameters but with coil elevated and angled away from the head)every day for ten consecutive days (5 days/week).
  Arms: Sham rTMS

SUMMARY:
The purpose of this study isto assess the efficacy of daily 10 sessions of rTMS over primary motor cortex in patients suffering from malignant neuropathic pain. Thirty four patients were divided randomly into 2 groups equally using closed envelops to undergo real (20 Hz, 10 second, 10 trains with inter-train interval 30 second with total pulses 2000, intensity 80% of motor threshold over hand area of motor cortex) or sham rTMS (same parameters but with coil elevated and angled away from the head)every day for ten consecutive days (5 days/week). Patients were evaluated using a verbal descriptor scale (VDS), visual analog scale (VAS), Leeds assessment of neuropathic symptoms and signs (LANSS) and Hamilton rating scale for depression (HAM-D) at baseline, after 1st, 5th, 10thtreatment session, and then 15 days and 1 month after the end of treatment. ic pain.

ELIGIBILITY:
Inclusion Criteria:

All patients within age group 18-65 years with malignant lateralized neuropathic pain resistant to medical treatment for at least 2 months or associated with significant adverse effects from medication were involved in this study.

Exclusion Criteria:

Patients with intracranial metallic devices Patients with pacemakers or any other device. Patients with recent myocardial ischemia, unstable angina Patients known to have history of epilepsy.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Neuropathic pain improvement | one month
  Reduction of neuropathic pain in patients with malignancy measured by VDS, VAS, LANSS.

SECONDARY OUTCOMES:
Reduction of depression manifestation | one month
  Measurement of depression by using (HAM-D) scale.